CLINICAL TRIAL: NCT07322809
Title: Association Between Postoperative Frailty Trajectories and One-Year Mortality in Older Surgical Patients: A Prospective Longitudinal Data Study
Brief Title: Postoperative Frailty Trajectories and One-Year Mortality in Older Surgical Patients
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yanhong Liu, Deputy Chief of administration, Anesthesiology, Chinese PLA General Hospital
Other Study IDs: PLAGH - FRAIL Trajectory
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Frailty in Older Adults; All Cause Mortality; Trajectory
Keywords: Frailty trajectory; older surgical patients; one-year mortality; latent class trajectory modeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A retrospective cohort study based on prospectively collected data.: Patients' frailty was assessed using the FRAIL scale at four time points: preoperatively and at 1, 3, and 6 months postoperatively. Patients were classified into distinct frailty trajectory groups using latent class trajectory modeling. The study examined the associations between frailty trajectories and one-year mortality and further identified independent factors associated with frailty trajectory membership.

SUMMARY:
Frailty is a key predictor of adverse outcomes in older surgical patients, yet its longitudinal evolution and potentially reversible nature remain underexplored in perioperative settings. This study aimed to characterize postoperative frailty trajectories in older patients and to examine their association with one-year mortality, as well as factors influencing trajectory group.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥65 years;
* Underwent elective non-cardiac, non-neurosurgical procedures;
* Completed standardized frailty assessments both preoperatively and postoperatively.

Exclusion Criteria:

* Severe dementia, language disorders, significant hearing or visual impairments, or coma;
* Cognitive function below the Mini-Mental State Examination (MMSE) thresholds (<18 for illiterate individuals, <21 for individuals with primary education, and <25 for individuals with secondary education or higher);
* Surgery performed under local anesthesia or monitored anesthesia care;
* Surgical duration ≤30 minutes;
* Missing data on postoperative complications or one-year mortality required for this study;
* Incomplete frailty assessments at 1, 3, and 6 months after surgery.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients' frailty was assessed using the FRAIL scale at four time points: preoperatively and at 1, 3, and 6 months postoperatively. Patients were classified into distinct frailty trajectory groups using latent class trajectory modeling. One-year all-cause mortality was ascertained through structured telephone follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 4417 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome was one-year all-cause mortality. | At the one-year postoperative follow-up.
  The primary outcome was one-year all-cause mortality, determined through structured telephone follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- 28 Fuxing Road, Haidian District, Beijin, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No